CLINICAL TRIAL: NCT05199740
Title: Assess the mtDNA Mutation Load in Mesoangioblasts of mtDNA Mutation Carriers
Brief Title: mtDNA Mutation Load Analysis in Mesoangioblasts
Acronym: MABS05
Status: Recruiting | Type: Observational
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Other Study IDs: NL78411.068.21
Record Dates: First submitted 2021-12-17; First posted 2022-01-20 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Mitochondrial Myopathies
MeSH Terms: conditions — Mitochondrial Myopathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — muscle derived cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mtDNA mutation carriers: Carriers of a pathogenic mtDNA mutation
  Interventions: Other: in vitro analysis

INTERVENTIONS:
Other: in vitro analysis — in vitro analysis of mesoangioblasts from mtDNA mutation carriers

SUMMARY:
Mitochondrial diseases caused by defects in oxidative phosphorylation (OXPHOS) due to heteroplasmic mitochondrial DNA (mtDNA) mutations are rare (frequency 1/5,000), but severe multi-system disorders. Clinical manifestations are highly variable, but predominantly affect energy demanding tissues, like brain and muscle. Myopathy is a common feature of mtDNA disorders, being present in more than 50% of the mtDNA mutation carriers, and seriously affects patients' general well-being and quality of life. Currently, no treatment is available for these patients, although the induction of muscle regeneration by exercise treatment has been shown to alleviate their myopathy. This implies that these patients can produce muscle fibres that perform better, most likely because the mutation load is lower. Mesoangioblasts (MABs) are myogenic precursors that have been recognized as a source for development of a systemic myogenic stem-cell therapy. Autologous MABs may be feasible for half of the mtDNA mutation carriers of 6 different mtDNA mutations, as their mtDNA mutation load in mesoangioblasts was (nearly) absent (<10%). However, there are many more mtDNA mutations in the 16.5kb mtDNA and the aim of this study is to determine the mtDNA mutation load in mesoangioblasts of other mtDNA mutation carriers and identify the patients or mutations for which this is a feasible approach.

DETAILED DESCRIPTION:
Rationale: Mitochondrial diseases caused by defects in oxidative phosphorylation (OXPHOS) due to heteroplasmic mitochondrial DNA (mtDNA) mutations are rare (frequency 1/5,000), but severe multi-system disorders. Clinical manifestations are highly variable, but predominantly affect energy demanding tissues, like brain and muscle. Myopathy is a common feature of mtDNA disorders, being present in more than 50% of the mtDNA mutation carriers, and seriously affects patients' general well-being and quality of life. Currently, no treatment is available for these patients, although the induction of muscle regeneration by exercise treatment has been shown to alleviate their myopathy. This implies that these patients can produce muscle fibres that perform better, most likely because the mutation load is lower. Mesoangioblasts (MABs) are myogenic precursors that have been recognized as a source for development of a systemic myogenic stem-cell therapy, and allogeneic transplantation has been successfully applied to mice and dogs with Duchenne muscular dystrophy. A subsequent phase I/II clinical study in boys with DMD demonstrated that donor MABs treatment was relatively safe, but did not result in clinical improvement, which can partly be attributed to the required use of immunosuppressive agents. The use of autologous MABs would circumvent this and a previous study of our group demonstrated that this is feasible for half of the mtDNA mutation carriers of 6 different mtDNA mutations, as their mtDNA mutation load in mesoangioblasts was (nearly) absent (<10%). However, there are many more mtDNA mutations in the 16.5kb mtDNA and the aim of this study is to determine the mtDNA mutation load in mesoangioblasts of other mtDNA mutation carriers and identify the patients or mutations for which this is a feasible approach.

Objective: The primary objectives of this project is to assess the mtDNA mutation load in mesoangioblasts of mtDNA mutation carriers and identify which patients display no/low (<10%) mtDNA mutation load in mesoangioblasts. Secondary objectives aim at determining the proliferation, myogenic differentiation and OXPHOS capacity of mesoangioblasts, their systemic inflammation status and assessment of the mtDNA mutation load in satellite cells.

Study design: Mono-centre observation study. Study population: 30 adult carriers of a heteroplasmic mtDNA point-mutation or large-scale mtDNA deletion (>2kb).

Intervention: From each participant, a 30mg skeletal muscle biopsy and a 20ml venous blood sample will be collected.

Main study parameters/endpoints: Assess the mtDNA mutation load in skeletal muscle derived mesoangioblasts.

ELIGIBILITY:
Inclusion Criteria all participants:

* Written informed consent
* Age: 18+
* Sex: male/female
* Carriers of a heteroplasmic mtDNA mutation load >20% in skeletal muscle or >1% in blood

Exclusion Criteria all participants:

* No informed consent
* Use of anti-coagulants, anti-thrombotics and other medication influencing coagulation
* Have a weekly alcohol intake of ≥ 35 units (men) or ≥ 24 units (women)
* Current history of drug abuse
* A history of strokes
* Significant concurrent illness
* Ongoing participation in other clinical trials that contain an intervention
* Major surgery within 4 weeks of the visit
* Pregnant or lactating women
* Patients unable and/or unwilling to comply with treatment and study instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the study, the following study population will be included: Adult males and females with a heteroplasmic mitochondrial mtDNA mutation identified in blood and/or skeletal muscle. Mitochondrial disorders due to a mtDNA mutation are very heterogeneous and carriers can present a variety of clinical symptoms and at varying age. The mtDNA mutation can be identified via diagnostic mtDNA analysis upon suspected or biochemically confirmed mitochondrial disease. Alternatively, given the maternal inheritance of the mtDNA, the mutation can be identified in (currently) unaffected siblings or children of a clinically affected mtDNA mutation carrier.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Assess mtDNA mutation load in mesoangioblasts | 1 day
  Isolate mesoangioblasts and quantify mtDNA mutation load using GeneScan analysis

SECONDARY OUTCOMES:
Assess level of systemic inflammation marker TNFa in blood plasma | 1 day
  TNFa measurement in plasma (pg/ml)
Assess level of systemic tissue damage marker CK in blood plasma | 1 day
  CK measurement in plasma (U/l)
Assess level of systemic inflammation marker IL-6 in blood plasma | 1 day
  IL-6 measurement in plasma (pg/ml)
Assess level of systemic inflammation marker SDF-1 in blood plasma | 1 day
  SDF-1 measurement in plasma (pg/ml)
Assess mitochondrial function in mesoangioblasts | 1 day
  Assess mtDNA copynumber and OXPHOS capacity in mesoangioblasts
Assess myogenic differentiation capacity of mesoangioblasts | 1 day
  Assess myogenic fusion index of mesoangioblasts isolated from a muscle biopsy
Assess mtDNA mutation load in satellite cells | 1 day
  Isolate satellite cells and quantify mtDNA mutation load using GeneScan analysis

CONTACTS AND LOCATIONS:
Overall Officials: Janneke Hoeijmakers, PhD, MD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No